CLINICAL TRIAL: NCT02775864
Title: Comparative Effectiveness of Adaptive Treatment Strategies for Schizophrenia
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Rutgers University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Scott Stroup, Professor, Columbia University
Other Study IDs: 7226
Record Dates: First submitted 2016-05-13; First posted 2016-05-18 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Antipsychotic Agents; Antidepressive Agents; Benzodiazepines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Antipsychotic: Individuals initiating treatment with an antipsychotic medication
  Interventions: Drug: Antipsychotic
- Antidepressant: Individuals initiating treatment with an antidepressant medication
  Interventions: Drug: Antidepressant
- Benzodiazepine: Individuals initiating treatment with a benzodiazepine
  Interventions: Drug: Benzodiazepine
- Mood stabilizer: Individuals initiating treatment with a mood stabilizer
  Interventions: Drug: Mood stabilizer

INTERVENTIONS:
Drug: Antipsychotic — New initiation of any antipsychotic medication
  Groups: Antipsychotic
Drug: Antidepressant — New initiation of any antidepressant medications
  Groups: Antidepressant
Drug: Benzodiazepine — New initiation of any benzodiazepine
  Groups: Benzodiazepine
Drug: Mood stabilizer — New initiation of lithium or any mood stabilizing anti-epileptic drug
  Groups: Mood stabilizer

SUMMARY:
The study is a retrospective cohort study of adults with schizophrenia that will compare outcomes of new users of alternative psychotropic medication strategies using 10 years of Medicaid data. The primary comparative effectiveness analyses will focus on subgroups of patients with schizophrenia facing common clinical situations.

DETAILED DESCRIPTION:
This retrospective cohort study will use data from national (45-state) Medicaid Analytic Extracts data (2001-2010). The cohort will consist of adults who are 18 to 64 years old and diagnosed with schizophrenia who initiate a new psychotropic medication after a period of stable antipsychotic treatment.

The eligibility criteria select a cohort of individuals diagnosed with schizophrenia, have received antipsychotic monotherapy prior to the index date, and are still experiencing problems for which a new psychotropic medication strategy was initiated. A 1-year period of eligibility prior to follow-up initiation ensures sufficient time to collect service use related covariates to characterize cohort members.

Five clinical subgroups will be defined based on the presence of psychiatric diagnoses during the 30 days prior to and inclusive of the treatment change under study (index date) and who have this same diagnostic code from more than one provider to increase the validity of the diagnostic groups. The subgroups will be defined by codes to capture 1) uncomplicated schizophrenia; 2) schizoaffective disorder; 3) depression; 4) mania; and 5) anxiety. These subgroups are defined to reflect the reason for the change in treatment.

Pharmacological treatment options for patients with schizophrenia who are nonresponsive to antipsychotic monotherapy will include (1) initiation of a second antipsychotic, (2) initiation of an antidepressant, (3) initiation of a mood stabilizer and (4) initiation of a benzodiazepine.

The primary effectiveness outcome will be time to psychiatric hospitalization. Secondary measures include time to index treatment discontinuation, time to introduction of another psychotropic medication, psychiatric emergency department visits, all-cause hospitalization, and death.

ELIGIBILITY:
Inclusion Criteria:

* The data source will be national (45-state) Medicaid Analytic Extracts data (2001-2010). The cohort will consist of adults who are 18 to 64 years old and diagnosed with schizophrenia who initiate a new psychotropic medication after a period of stable antipsychotic treatment.

  * Schizophrenia will be defined as ≥2 outpatient claims or ≥1 inpatient claim for schizophrenia [ICD-9-CM: 295] during 365 days of consecutive Medicaid enrollment immediately prior to the index date. Stable antipsychotic monotherapy will be defined by filled prescriptions for only one second-generation antipsychotic, and no other psychotropics, for ≥ 90 days immediately preceding the start of the index medication (t0). After the ≥90 days of stable treatment with a single second-generation antipsychotic, study patients will have had a change in therapy defined as (1) addition of a second antipsychotic or (2) addition of a different psychotropic drug class (antidepressant, mood stabilizer, or benzodiazepine). To ensure the patients are in active treatment there must be an active supply of antipsychotic medication on t0.

Exclusion Criteria:

* Medicare recipients
* Patients receiving clozapine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults diagnosed with schizophrenia who are taking only a single antipsychotic medication who initiate treatment with an additional psychotropic medication.
Sampling Method: Non-Probability Sample
Enrollment: 81921 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer
Started | 26014 | 31117 | 11941 | 12849
Completed | 22772 | 26218 | 10081 | 10765
Not Completed | 3242 | 4899 | 1860 | 2084
Not completed — Data ended end of 2010 | 1764 | 2880 | 1140 | 1194
Not completed — Medicaid eligibility discontinued | 1478 | 2019 | 720 | 890

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer | Total
Number analyzed (Participants) | 26014 | 31117 | 11941 | 12849 | 81921
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.5) | 40.5 (12.4) | 40.5 (12.5) | 40.3 (12.5) | 40.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11914 | 14283 | 5553 | 5975 | 37725
  Male | 14100 | 16834 | 6388 | 6874 | 44196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 9645 | 10998 | 5186 | 4261 | 30090
  Black, non-Hispanic | 10371 | 12459 | 3731 | 5465 | 32026
  Hispanic or Latino | 2517 | 3196 | 1159 | 1263 | 8135
  Asian | 645 | 461 | 252 | 237 | 1595
  Hawaiian or Pacific Islander | 782 | 744 | 339 | 287 | 2152
  Native American or Alaskan Native | 240 | 305 | 104 | 87 | 736
  More than one race | 51 | 67 | 19 | 26 | 163
  Unknown | 2763 | 2787 | 1152 | 1223 | 7925

OUTCOME MEASURES:

1. Primary Outcome: Psychiatric Hospitalization
Description: Number of participants hospitalized for a mental health reason
Time Frame: One year
Measure: Count of Participants; unit: Participants
Groups:
- Antipsychotic: Individuals initiating treatment with another second-generation antipsychotic medication (other than clozapine
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer
Number analyzed (Participants) | 26014 | 31117 | 11941 | 12849
Participants | 4965 | 5247 | 2385 | 3093

2. Secondary Outcome: Emergency Department Visit for Mental Health Reason
Description: Number of Participants with an Emergency Department visit for mental health reason
Time Frame: One year
Measure: Count of Participants; unit: Participants
Groups:
- Antipsychotic: Individuals initiating treatment with another second-generation antipsychotic medication (other than clozapine)
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer
Number analyzed (Participants) | 26014 | 31117 | 11941 | 12849
Participants | 5505 | 6508 | 2930 | 3429

3. Secondary Outcome: Death
Description: Participants who died
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer
Number analyzed (Participants) | 26014 | 31117 | 11941 | 12849
Participants | 259 | 327 | 204 | 161

ADVERSE EVENTS:
Time Frame: 365 days
Arm/Group | Antipsychotic | Antidepressant | Benzodiazepine | Mood Stabilizer
All-Cause Mortality (participants affected / at risk) | 259/26014 | 327/31117 | 204/11941 | 161/12849
Serious Adverse Events (participants affected / at risk) | 67/26014 | 102/31117 | 43/11941 | 41/12849
Other Adverse Events (participants affected / at risk) | 967/21738 | 1004/26062 | 424/9764 | 423/10564
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antipsychotic (N=26014) | Antidepressant (N=31117) | Benzodiazepine (N=11941) | Mood Stabilizer (N=12849)
Admission for Cardiovascular Disease (Cardiac disorders) | 67 | 102 | 43 | 41 — Defined by first listed diagnosis of acute myocardial infarction (AMI) (ICD-9-CM: 410) or stroke (430-438, except 435) on inpatient claims.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antipsychotic (N=21738) | Antidepressant (N=26062) | Benzodiazepine (N=9764) | Mood Stabilizer (N=10564)
Incident cases of diabetes mellitus (Endocrine disorders) | 967 (967) | 1004 (1004) | 424 (424) | 423 (423)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT02775864/Prot_SAP_000.pdf